CLINICAL TRIAL: NCT01648673
Title: Pilot Evaluation of the Janssen Healthcare Innovation Integrated Cardiovascular Rehabilitation Management Platform (JHI PLATFORM).
Brief Title: Pilot Evaluation of the JHI Platform
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Steven J. Keteyian, Program Director, Henry Ford Health System
Other Study IDs: HFHS-JHI Platform
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Cardiac Rehabilitation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose of this pilot study is to evaluate an impact of JHI CR Platform on patient referral, recruitment and retention rates and overall patient satisfaction in cardiovascular rehabilitation programs at the HFHS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 years old (inclusive) and older
* Recent hospitalization at HFHS Main Campus hospital with one of the following diagnosis
* Stable angina with medical management
* Myocardial infarction (MI)/Acute coronary syndrome
* Percutaneous Coronary Intervention (PCI)
* Coronary Artery Bypass Graft (CABG) surgery
* Heart valve surgical repair or replacement
* Patients must be attending outpatient CR program at the HFHS Detroit location.
* Willingness to participate in the study and follow study requirements
* Willingness to respond to several surveys at the baseline and periodically during the study

Exclusion Criteria:

* Active substance abuse per medical record
* Unstable psychiatric condition
* Inability to exercise
* Unstable medical condition that would prevent safe and regular exercise training
* Uncorrected Severe Aortic Stenosis or Severe Mitral Stenosis
* Inpatient referring physician feels that exercise in contra-indicated due to safety reasons or is ill advised due to other patient specific factors
* LVAD, Heart Transplant. Although these patients qualify for CR, HFHS is not recruiting them due to difficulty in coordinating with surgical patients and their providers. In addition, there may also be surgical issues (infection, wound dehiscence, bone healing etc) that may reasonably interfere with exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiology services.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Patient referral, recruitment and retention rates and overall patient satisfaction. | Beginning, middle, and end of participation.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Keteyian, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States